CLINICAL TRIAL: NCT01806246
Title: An Integrative Approach Based Psychoeducation, Heart Rate Variability Coherence Biofeedback and Elements of, Pacing Cognitive Behavior Therapy
Brief Title: A Rehabilitation Program for Adolescents With Chronic Fatigue Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/2159
Record Dates: First submitted 2013-03-01; First posted 2013-03-07 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Fatigue Syndrome
Keywords: rehabilitation; adolescent; heart rate variability biofeedback; psychoeducation
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- integrative rehabilitation program (Experimental): 28 sessions during 12 months with focus on psychoeducation, activity planning, and thoughts and feelings connected to having a serious chronic disease. From week 13 to week 32 a training programme aiming at balancing heart rate variability.
  Interventions: Behavioral: integrative rehabilitation program

INTERVENTIONS:
Behavioral: integrative rehabilitation program

SUMMARY:
The aim of the programme is to develop a treatment model for adolescents with Chronic Fatigue Syndrome. The program consists of 4 elements lasting for 12 months, psychoeducation reflecting the current knowledge about the disease, Heart Rate Variability Coherence Biofeedback, pacing and activity planning and some principles of cognitive behaviour therapy. The study is designed as a Single-Case study including 10- 15 participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet the diagnostic criteria of chronic fatigue syndrome
* Clinically evaluated, exclude any disease that can explain the chronic fatigue;
* Diagnosed and evaluated within the health region, Central Norway
* With written consent form signed by themselves and their parents.

Exclusion Criteria:

* serious comorbidity such as anorexia, psychosis
* serious depression

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2013-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
fatigue change | baseline and 52 weeks
  assessed by Fatigue Severity Scale
quality of life change | baseline and 52 weeks
  assessed by Inventory of Life Quality for Children and Adolescents

SECONDARY OUTCOMES:
mood change | baseline and 52 weeks
  assessed by Mood and Feelings Questionnaire
change in heart rate variability | baseline and 52 weeks
school attendance change | baseline and 52 weeks
general health change | baseline and 52 weeks
  General Health Questionnaire (GHQ-12)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jozefiak, md phd, Study Director — St. Olavs Hospital
Locations (1):
- Dept Child and Adolescent Psychiatry, St Olavs Hospital, Trondheim, Norway